CLINICAL TRIAL: NCT00276432
Title: Diagnosis and Treatment of Acute Coronary Syndrome in the Emergency Department- The Impact of Rapid Bedside cTnl on Outcome.
Brief Title: Diagnosis and Treatment of Acute Coronary Syndrome in the ED & the Impact of Rapid Bedside cTnl on Outcome.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Abbott (Industry); University of Cincinnati (Other); Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 637-05
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Unstable Angina; Non-ST-Elevation Myocardial Infarction
MeSH Terms: conditions — Angina, Unstable; Non-ST Elevated Myocardial Infarction

INTERVENTIONS:
Device: iSTAT point of care analyzer

SUMMARY:
The primary outcome in this study will be time to discharge for low-risk patients and therapeutic turnaround time for patients with NSTEMI or unstable angina.

DETAILED DESCRIPTION:
Phase IV prospective, randomized (1:1), parallel-group trial utilizing concurrent controls. Assess the reduction in time taken to dispostion or discharge patients. Assess the ability of POC testing to satisfy guidelines for a 30 minute turn around time of results. Assess and differences in clinical decision-making for other diagnostic procedures including nuclear imaging, echo, and stress treadmill, disposition from the ED, time to catherterization lab, PCI, and CafBG based on the cardiac troponinn results from the bedside analyzer and the central lab instrument.Assess the difference for in-hospital and 30 day post hospital discharge cardiac events including all-cause and cardiac-specific deaths, CHF, cardiomyopathy, and atrial and ventricular arrhythmia, beween the bedside analyzer and the central lab instrument. Assess the differences in hospital care costs for the hospitalization period, and assess direct medical and indirect productivity costs in the 30 day post hospital discharge period to patients who are diagnosed, using the bedside cTnl test and the central lab cTn tests, and subsequently treated as per the guidelines.

ELIGIBILITY:
Patient must be 21 years old or older with chest pain or other symptoms that lead to drawing cardiac biomarkers.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to discharge for low-risk patients
Therapeutic turnaround time for patients with NSTEMI or unstable angina

CONTACTS AND LOCATIONS:
Overall Officials: Wyatt W. Decker, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States